CLINICAL TRIAL: NCT06990490
Title: A Novel Endoscopy-Guided Airway Management Strategy for Lateral Decubitus Endoscopic Procedures
Brief Title: Application of Lateral Position Digestive Endoscopy-Guided Endotracheal Intubation in Anesthesia for Endoscopic Diagnosis and Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Changlong Qiao (Other)
Responsible Party: Sponsor-Investigator, Changlong Qiao, Attending Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(028)
Record Dates: First submitted 2025-05-10; First posted 2025-05-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Endotracheal Intubation; Gastrointestinal Endoscopy; Airway Management; Lateral Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This case series study evaluated whether placing a breathing tube using a camera (gastrointestinal endoscope) is safe and effective for patients lying on their left side during stomach and intestine exams under anesthesia. The main questions were:

How often does the tube placement work on the first try? How long does it take to place the tube? Are there any safety issues, like injuries or breathing problems?

Researchers enrolled 40 adults needing anesthesia for stomach/intestine exams. All participants had the breathing tube placed while lying on their left side using the camera-guided method. The steps included:

Positioning the patient on their left side with head/neck support. Inserting a lubricated camera through the mouth to view the throat. Placing the breathing tube into the windpipe under direct camera view.

The method avoided the risks of moving anesthetized patients from their back to the side. It may reduce risks linked to repositioning patients during surgery. Future studies with more participants and different medical teams are needed to confirm these results.

ELIGIBILITY:
Inclusion Criteria:

* The study population comprised individuals requiring endotracheal intubation during elective gastrointestinal endoscopy in the left lateral position

Exclusion Criteria:

* Patients who declined informed consent were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This investigation was a case series study conducted in The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital between February 2025 and March 2025. The study population comprised individuals requiring endotracheal intubation during elective gastrointestinal endoscopy in the left lateral position. Patients who declined informed consent were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of the first intubation attempt and intubation time (from endoscope insertion to tube connection) | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China